CLINICAL TRIAL: NCT04605718
Title: A Randomized, Sponsor-Open, Adaptive, Single- And Multiple-Ascending Dose, Placebo-Controlled Study To Investigate The Safety, Tolerability, And Pharmacokinetics Of RO7223280 Following Intravenous Administration In Healthy Participants
Brief Title: A Study To Investigate The Safety, Tolerability And Pharmacokinetics (PK) Of RO7223280 Following Intravenous Administration In Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BP41732
Record Dates: First submitted 2020-10-23; First posted 2020-10-28 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (SAD) (Experimental): Due to mandatory sentinel dosing, participants will be divided into two groups: 2 participants will be dosed on one day (sentinel group with 1 on active treatment and 1 on placebo) and remaining participants of the dose cohort (randomized as 5 on active treatment and 1 on placebo) at the earliest 24 hours after the first dosing occasion.
  Interventions: Drug: RO7223280
- Part 2 (MAD) (Experimental): In each dose cohort, a minimum of 4 participants and a maximum of 12 participants will receive either multiple IV doses of RO72232809 or placebo once-daily for 10 days (3:1 ratio of active:placebo treatment).
  Interventions: Drug: RO7223280
- Part 3 (Elderly) (Experimental): In this cohort, a minimum of 4 participants and a maximum of 12 participants will receive a single IV dose of RO7223280 or placebo (3:1 ratio of active:placebo treatment).
  Interventions: Drug: RO7223280

INTERVENTIONS:
Drug: RO7223280 — For Part 1 (SAD) and Part 2 (MAD), RO7223280 will be administered by intravenous (IV) infusion at escalating doses from 10mg to 4800mg, as per the dosing schedules described above. These are putative doses and the maximum daily dose that must not be exceeded is 5000mg. For Part 3 (Elderly), RO7223280 will be administer as one single IV dose of 300 mg.

SUMMARY:
The Study consists of 3 Parts: Part 1 (Single Ascending Dose/SAD), Part 2 (Multiple Ascending Dose/MAD), and Part 3 (Elderly). Part 1 will investigate the safety, tolerability and PK of single-ascending intravenous (IV) doses of RO7223280 in healthy participants. Part 2 will investigate the safety, tolerability and PK of multiple-ascending IV doses of RO7223280 in healthy participants. Part 2 will start after the initial completion of Part 1 (SAD). Progression from Part 1 to Part 2 will be based on a satisfactory review of all available safety, tolerability, and PK data by the Investigator and the Sponsor from Part 1. The starting dose for Part 2 will be administered as 1-hour IV infusion; as it has been established on the basis of all available safety, tolerability, and PK data in Part 1 (SAD). Part 3 will investigate the safety, tolerability and PK of a single IV dose of RO7223280 in healthy elderly participants. A single IV dose of RO7223280 administered over 1 hour was selected, within the range of previously explored doses in Part 1 (SAD).

ELIGIBILITY:
Inclusion Criteria:

* Parts 1 (SAD) and 2 (MAD): 18 to 64 years of age, inclusive. Part 3 (Elderly): 65 years of age and older
* Healthy participants in Part 1 (SAD) and Part 2 (MAD). Health status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, serology, coagulation, and urinalysis. Healthy participants in Part 3 (Elderly). Participants must be in reasonably good health as determined by the Investigator based on medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology,blood chemistry, serology, coagulation, and urinalysis. Participants with mild, chronic, stable disease (e.g., controlled hypertension, controlled diabetes mellitus) may be enrolled if deemed medically prudent by the Investigator.
* In Part 1 (SAD) and Part 2 (MAD) participants must weigh at least 50 kg and must have a body mass index (BMI) within the range of 18 to 32 kg/m^2 (inclusive). In Part 3 (Elderly), participants must weigh at least 50 kg with no restrictions regarding the BMI.
* During the treatment period and for at least 90 days after the final dose of RO7223280 or placebo, male participants (whether surgically sterilized or not) agree to remain abstinent (refrain from heterosexual intercourse), use contraceptive measures and refrain from donating sperm at least 90 days after last dose.

Exclusion Criteria:

* For Part 1 (SAD) and Part 2 (MAD), history of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardiovascular, endocrinological, hematological or allergic disease, metabolic disorder, cancer, or cirrhosis.For Part 3 (elderly), participants must be in reasonably good health as determined by the Investigator based on a detailed medical history. Participants with mild, chronic, stable disease and on stable medication may be enrolled if deemed medically prudent by the Investigator.
* In Part 1 (SAD) and Part 2 (MAD), use of glucocorticoids and other immunosuppressive medications is prohibited within 30 days (or within 5 times the elimination half-life, whichever is longer), prior to Day 1. In Part 3 (Elderly Cohort), the systemic use of glucocorticoids and other immunosuppressive medications is prohibited within 30 days (or within 5 times the elimination half-life, whichever is longer), prior to Day 1.
* Participation in an investigational drug medicinal product or medical device study within 30 days prior to screening or within 5 times the elimination half-life if known, whichever is longer.
* In Part 1 (SAD) and Part 2 (MAD), confirmed (based on the average of 3 consecutive measurements) systolic blood pressure (SBP) greater than 140 or less than 90 mmHg, and diastolic blood pressure (DBP) greater than 90 or less than 50 mmHg at screening. In Part 3 (Elderly), confirmed (based on the average of 3 consecutive measurements) systolic blood pressure (SBP) greater than 160 or less than 80 mmHg, and diastolic blood pressure (DBP) greater than 90 or less than 40 mmHg at screening.
* Confirmed (based on the average of 3 consecutive measurements) resting pulse greater than 100 bpm or less than 40 bpm at screening.
* Positive for HIV or Hepatitis B/C infections.
* Donation of blood or blood products for transfusion over 500 mL within 3 months prior to first study drug administration and for the duration of the study.
* Any clinically significant history of hypersensitivity or allergic reactions, either spontaneous or following study drug administration, or from exposure to food or environmental agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to 19 months

SECONDARY OUTCOMES:
Plasma Concentrations of RO7223280 at specified timepoints | Up to 19 months
Urine Concentrations of RO7223280 at specified timepoints | Up to 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Covance Clinical Research Unit, Inc, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).